CLINICAL TRIAL: NCT01878708
Title: A Pilot Study of Oncaspar® + Dexamethasone in Patients With Relapsed or Refractory T-Cell Lymphoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Leadiant Biosciences, Inc. (Industry)
Responsible Party: Principal Investigator, Philippe Armand, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-165
Record Dates: First submitted 2013-05-23; First posted 2013-06-17 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: T-Cell Lymphoma; Relapsed T-Cell Lymphoma; Refractory T-Cell Lymphoma
Keywords: T-Cell Lymphoma; Relapsed T-Cell Lymphoma; Refractory T-Cell Lymphoma; Oncaspar®; PEG-L-asparaginase and dexamethasone
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — pegaspargase; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PEG-L-asparaginase/Dexamethasone (Experimental): Patients will receive Oncaspar® (PEG-asparaginase) at a dose of 2,000 IU/m2 administered intramuscularly on day 3 of each 3 week cycle, with dexamethasone 40mg given orally on days 1-4.
  Interventions: Drug: PEG-L-asparaginase; Drug: Dexamethasone acetate

INTERVENTIONS:
Drug: PEG-L-asparaginase
  Other Names: Oncaspar; PEG-asparaginase
Drug: Dexamethasone acetate — -dexamethasone 40mg daily for 4 days with every cycle.

SUMMARY:
This is an open-label, single-arm pilot study of Oncaspar® with dexamethasone for patients with relapsed or refractory peripheral T-cell lymphoma (PTCL), excluding extranodal NK/T cell lymphoma (ENKTL). Patients will receive up to 8 courses of treatment.

DETAILED DESCRIPTION:
This is an open-label, investigator-initiated, single-arm pilot study. Patients with relapsed or refractory (R/R) peripheral T-cell lymphoma (PTCL) will receive Oncaspar® every 3 weeks up to a maximum of 8 courses or until disease progression or unacceptable toxicity. They will also receive dexamethasone 40mg daily for 4 days with every cycle. They will be restaged after 2 courses (6 weeks) and after 8 courses (24 weeks).

Both Oncaspar and dexamethasone have been used together to treat ALL and ENKTL, which is another subtype of T cell lymphoma. The combination may provide a collaborative attack against the cancer cell; moreover, the dexamethasone could also prevent some of the side effects of Oncaspar; especially allergic reactions. This study will test these two drugs together to determine if they are an effective treatment for T-Cell Lymphoma. Each drug is commercially available to the drug market.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria on screening examination to be eligible to participate in the study:
* Patients must have histologically confirmed peripheral T-cell lymphoma, with the diagnostic specimen reviewed at one of the DFHCC hematopathology laboratories. Eligible histologies include:
* PTCL-NOS
* Systemic T cell/null anaplastic large cell lymphoma (ALCL), regardless of Alk status
* Angioimmunoblastic T-cell lymphoma (AITL)
* Hepatosplenic (alpha-beta or gamma-delta) lymphoma (HSL)
* Enteropathy-associated T-cell lymphoma (EATL)
* Adult T-cell leukemia/lymphoma (ATLL), lymphomatous subtype
* Subcutaneous panniculitis-like T-cell lymphoma
* T-cell Prolymphocytic Leukemia (T-PLL)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan
* Patients must have relapsed or progressed after at least 1 prior course of anti-lymphoma therapy.
* Age 18-65 years.
* ECOG performance status <2 (see Appendix A).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Patients with cutaneous disease only are not eligible.
* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier to grade 1 or below (unless approved by the Study Chair).
* Patients may not be receiving any other study agents at the time of first treatment.
* History of treatment with an asparaginase agent.
* Patients with a history of alcohol abuse, or patients unwilling or unable to remain completely abstinent of alcohol during the study period.
* Hepatitis B or C seropositivity (except for hepatitis B with negative surface antigen and hepatitis B viral load).
* Total bilirubin > institutional upper limit of normal (ULN), unless due to hemolysis or Gilbert's disease).
* AST/ALT ≥ 3 x ULN.
* History of pancreatitis, or amylase > ULN or lipase > ULN.
* History of thromboembolic disease.
* Grade 2 or above neuropathy.
* Diabetes mellitus, unless it is type II diabetes adequately controlled with anti-diabetic agents (A1c < 7).
* History of CNS hemorrhage or thrombosis. Patients with a history of CNS lymphomatous involvement are eligible only if their CNS disease is in remission at the time of study entry.
* Uncontrolled intercurrent illness including, but not limited to uncontrolled active infection, symptomatic congestive heart failure (New York Hospital Association (NYHA) class II-IV, resulting in at least slight limitation of activity), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Inability to provide informed consent
* Pregnancy or lactation.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* HIV-positive individuals on combination antiretroviral therapy are ineligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete + partial response) in evaluable patients. | 24 weeks

SECONDARY OUTCOMES:
Duration of response for patients with PR or CR | 24 weeks
Grade 2 and above attributable toxicity of treatment. | 24 weeks
Progression-free survival. | 1 year
  This will be assessed in both evaluable patients and in responders.
Complete remission (CR) rate. | 24 weeks
  This will be assessed both in the intent-to-treat and in the evaluable populations.
Partial remission (PR) rate. | 24 weeks
  This will be assessed both in the intent-to-treat and in the evaluable populations.
The stable disease (SD) rates in this population and in the intent-to-treat population | 24 weeks
Progressive disease (PD) rate. | 24 weeks
  This will be assessed both in the intent-to-treat and in the evaluable populations.
Stable disease (SD) rate. | 24 weeks
  This will be assessed both in the intent-to-treat and in the evaluable populations.
Overall survival | 1 year
  This will be assessed in both evaluable patients and in responders.

CONTACTS AND LOCATIONS:
Overall Officials: Phillippe Armand, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No